CLINICAL TRIAL: NCT05416918
Title: Assessing the Clinical Value of Metagenomics Sequencing for the Diagnosis and Treatment of Neonatal Sepsis: a Multicenter Prospective Observational Study
Brief Title: Clinical Value of Metagenomic Sequencing in Neonatal Sepsis
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Quanzhou Women's and Children's Hospital (Unknown); Shengjing Hospital (Other); Jiangxi Maternal and Child Health Hospital (Other); Northwest Women's and Children's Hospital, Xi'an, Shaanxi (Other); Nanjing Maternity and Child Health Care Hospital (Other); The First Hospital of Jilin University (Other); Hunan Children's Hospital (Other Government); Henan Provincial People's Hospital (Other); Tianjin Central Hospital of Gynecology Obstetrics (Other); Jiangxi Children's Hospital (Unknown); Maternal and Child Health Hospital of Guangxi Zhuang Autonomous Region (Other); Xinjiang Children's Hospital (Unknown); Shenzhen Maternity and Child Healthcare Hospital (Unknown); Children's Hospital of Nanjing Medical University (Other); Gansu Provincial Maternal and Child Health Care Hospital (Other); Kunming Children's Hospital (Other); Fujian Provincial Maternity and Children (Unknown); Zhuhai Women and Children's Hospital (Unknown); Xiamen Children's Hospital (Other); Children's Hospital Affiliated to Shandong University (Unknown); Henan Maternal and Child Health Care Hospital (Unknown); Wuhan Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CHFudanU_NNICU18
Record Dates: First submitted 2022-06-02; First posted 2022-06-14 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Neonatal Sepsis
Keywords: Neonatal Sepsis; Metagenomics; High-Throughput Nucleotide Sequencing
MeSH Terms: conditions — Neonatal Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — At the same time of sending conventional blood culture or cerebrospinal fluid culture, 2ml of blood and 1ml of cerebrospinal fluid were collected additionally.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aimed to enroll 2000 neonatal patients with suspected sepsis or clinical diagnosed sepsis. These patients will undergo both conventional methods and metagenomics sequencing to detect the pathogenic microorganisms of sepsis. The purpose of this study was to assess the clinical value of metagenomics sequencing for the diagnosis and treatment of neonatal sepsis.

DETAILED DESCRIPTION:
Infectious diseases remain leading causes of mortality and morbidity in children. Rapid and accurate diagnosis of infectious diseases in children is important for developing an effective treatment and management strategy. However, the current diagnosis of infectious agents mainly depends on culture and molecular testing. Both of the methods either has long turnaround times or narrow detection range. Metagenome next generation sequencing (mNGS) has been applied to the diagnosis of central nervous system infection, lower respiratory tract infection and sepsis, which showed high positive rate, short turnaround time. As a multi-center prospective observational clinical study, the study intends to enroll 2000 suspected neonatal sepsis cases from multiple centers. Culture, classical PCR and mNGS were performed simultaneously. This study is one of the few multi-center studies in China to evaluate the value of mNGS in the diagnosis and treatment of neonatal sepsis, and will provide representative data for the distribution characteristics of pathogen spectrum of children in the real world and the clinical diagnosis and treatment value of mNGS.

ELIGIBILITY:
Inclusion Criteria:

* Neonates with suspected early-onset sepsis or late-onset sepsis;
* Neonates diagnosed with clinical sepsis.

Exclusion Criteria:

* Died before the results of conventional methods test or metagenomics test were obtained;
* Suffering from diseases of the blood system;
* Suffering from malignant tumor;
* Birth defects, congenital heart disease or autoimmune disease.

Ages: 0 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study focuses on neonates with primary clinical diagnosis of sepsis.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance of metagenomics sequencing | From the date of first samples enrolled until the last samples detected, up to 2 years.
  The diagnostic performance of metagenomics sequencing for neonatal sepsis was evaluated by calculating sensitivity and specificity. Sensitivity = mNGS positive samples/ reference standard methods positive samples; Specificity = mNGS negative samples/ reference standard methods negative samples.

SECONDARY OUTCOMES:
Clinical impact of metagenomics sequencing | From the date of first samples enrolled until the last samples detected, up to 2 years.
  Clinical impact of metagenomics sequencing was evaluated by calculating the positive impact rate, negative impact rate and no impact rate. Positive impact rate = positive impact cases/ total cases; negative impact rate = negative impact cases/ total cases; no impact rate = no impact cases/ total cases. Clinical impact was assessed according to predefined objective grading criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Wenhao Zhou, Doctor, Study Chair — Children's Hospital of Fudan University
Locations (1):
- Children Hospital of Fudan University, Shanghai, China